CLINICAL TRIAL: NCT01701440
Title: Radiofrequency Magnetic Induction Device for Use In Dermatologic Procedures for the Non-Invasive Treatment of Wrinkles and Rhytides
Brief Title: Efficacy Study for Magnetic Induction to Treat Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rocky Mountain Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0310-0017
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Wrinkles and Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Biofusionary Bebe

SUMMARY:
In this study we propose to test the Biofusionary Bebe in order to reduce skin laxity and improve contour and cosmesis.

ELIGIBILITY:
The inclusion criteria for the study are:

* Male or female 21 to 65 years old,
* Clinically appreciable skin laxity on the abdomen (including flank), face, neck, hips, thighs, upper arms & buttocks as determined by the study investigator,
* For females, post-menopausal, surgically sterilized, or using a medically accepted form of birth control for at least 3 months prior to the study,
* Apparently healthy,
* Informed consent signed by the subject.

Exclusion Criteria:

The exclusion criteria for the study are:

* History of skin hypersensitivity,
* Current skin disorder (e.g. keloid scarring) or infection (e.g., herpes simplex) in the treatment area,
* Subjects with pacemakers, internal defibrillators or electronically, magnetically, and mechanically activated implants,
* Subjects with implanted medical prostheses (such as clips, pins or plates) proximal to the treatment site,
* The current or recent use (within the past 12 months) of isotretinoin,
* Pregnancy,
* Infectious diseases (such as HIV) present,
* Are a tobacco smoker,
* Insulin dependent diabetic subjects,
* Oxygen dependent subjects,
* Subjects with severe chronic illness, scleroderma, or lupus,
* Subjects with open sores or scars in the treatment region, or
* Subjects with ischemia in the treatment region.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in cosmesis | 1 month
  Improvement in cosmesis will be assessed by scoring photographs taken before and 1 month after treatment. Circumference changes will be measured and compared

SECONDARY OUTCOMES:
Improvement in cosmesis | 3 months
  Improvement in cosmesis will be assessed by scoring photographs taken before and at 3 months after treatment. Circumference changes will be measured and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Garden, MD, Principal Investigator — Physicians Laser and Dermatology Institute of Chicago
Locations (1):
- Physicians Laser and Dermatolgy Institute of Chicago,LLC, Chicago, Illinois, United States